CLINICAL TRIAL: NCT04809025
Title: Comparation of Endoscopic Biopsy and Postoperative Specimen for the Molecular Diagnosis of Gastric Cancer
Acronym: EBPS
Status: Recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Dazhi Xu, professor, Fudan University
Other Study IDs: EBPS
Record Dates: First submitted 2021-03-19; First posted 2021-03-22 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Stomach Neoplasms; Endoscopy; Biopsy; Pathology
Keywords: Stomach Neoplasms; Endoscopy; Biopsy; Pathology
MeSH Terms: conditions — Stomach Neoplasms | interventions — Endoscopy; Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — preoperative endoscopic biopsy specimens and postoperative specimen of gastric tumors
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- the pathology of endoscopic biopsy: The histological type, histological grade, LAUREN type, HER-2 expression, MSI/dMMR status, and EBV status of gastric cancer testing on endoscopic biopsies
  Interventions: Device: endoscopy
- the pathology of surgical resection specimen: The histological type, histological grade, LAUREN type, HER-2 expression, MSI/dMMR status, and EBV status of gastric cancer testing on surgical resection specimens
  Interventions: Procedure: Surgery

INTERVENTIONS:
Device: endoscopy — gastroscope
  Groups: the pathology of endoscopic biopsy
Procedure: Surgery — radical gastrectomy
  Groups: the pathology of surgical resection specimen

SUMMARY:
This study aims to test the hypothesis that the diagnosis for histological type, histological grade, LAUREN type, HER-2 expression, MSI/dMMR status, and EBV status in gastric cancer is at least as reliable when performed on endoscopic biopsy specimens as on surgical resection specimens.

DETAILED DESCRIPTION:
Most institutions currently diagnose gastric cancer on endoscopic biopsy specimens but use surgical resection specimens for histological type, histological grade, LAUREN type, HER-2 expression, MSI/dMMR status and EBV status testing. However, gastric cancers treated with neoadjuvant chemoradiotherapy/chemotherapy may undergo a complete pathological response (pCR), with no residual tumors available for testing, and neoadjuvant chemoradiotherapy/chemotherapy may alter the HER-2 expression, MSI/dMMR status and EBV status of the gastric cancer in some instances. Importantly, testing histological type, histological grade, LAUREN type, HER-2 expression, MSI/dMMR status and EBV status of gastric cancer on endoscopic biopsy material could be initiated preoperatively, allowing resultant genetic information to be used in consultation with the patient to inform treatment decisions. Therefore, the preoperative endoscopic biopsy may be a source of suitable and reliable testing material. This study aims to investigate the correlation between histological type, histological grade, LAUREN type, HER-2 expression, MSI/dMMR status, and EBV status in preoperative endoscopic biopsy specimens and their corresponding surgical resection specimens and ascertain whether endoscopic biopsy specimen is a valid and reliable testing material for determining the histological type, histological grade, LAUREN type, HER-2 expression, MSI/dMMR status and EBV status of gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Lower age limit of research subjects 18 years old and upper age limit of 75 years old.
2. Histologically proven primary gastric adenocarcinoma (Diagnostic biopsies must be collected within 12 months prior to enrollment).
3. Written informed consent from the patient.
4. Patients planned for radical R0 gastrectomy.

Exclusion Criteria:

1. Female in pregnancy or lactation.
2. Patients with gastric cancer who can not undergo tumor resection
3. Suffering from other serious diseases, including cardiovascular, respiratory, kidney, or liver disease, complicated by poorly controlled hypertension, diabetes, mental disorders or diseases.
4. Patients with poor compliance or considered to be poor compliance.
5. Patients received any anticancer drugs, biotherapy, radiotherapy or immunotherapy within 4 weeks before or after enrollment.
6. Patients after organ transplantation, long-term need to take immunosuppressants, autoimmune diseases.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Treatment-naive gastric cancer patients
Sampling Method: Probability Sample
Enrollment: 510 (Estimated)
Dates: Start 2021-05-24 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy | 2-year
  The primary outcome of this trial is to investigate the correlation between histological type, histological grade, LAUREN type, HER-2 expression, MSI/dMMR status and EBV status in pretreatment endoscopic biopsy specimens and their corresponding surgical resection specimens

SECONDARY OUTCOMES:
The proportion of incomplete molecular pathology detection | 2-year
  incomplete molecular pathology detection defined as endoscopic biopsy specimens and surgical resection specimens from which the definitive histological type, histological grade, LAUREN type, HER-2 expression, MSI/dMMR status and EBV status diagnosis cannot be rendered by the pathologist
Procedure duration | 2-year
  The total length of time for the diagnosis of histological type, histological grade, LAUREN type, HER-2 expression, MSI/dMMR status and EBV status performed on endoscopic biopsy specimens and surgical resection specimens will be documented(days).

CONTACTS AND LOCATIONS:
Overall Officials: Dazhi Xu, PHD, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China